CLINICAL TRIAL: NCT03528629
Title: A Phase 1 Open-label Study of IMAB362 in Japanese Subjects With Locally Advanced or Metastatic Gastric or Gastro-esophageal Junction (GEJ) Adenocarcinoma
Brief Title: A Study of IMAB362 in Japanese Subjects With Locally Advanced or Metastatic Gastric or Gastro-esophageal Junction (GEJ) Adenocarcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 8951-CL-0104; jRCT2080223901 (Other: jRCT)
Record Dates: First submitted 2018-05-06; First posted 2018-05-18 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Gastric Cancer; Gastro-esophageal Junction (GEJ) Cancer
Keywords: zolbetuximab; IMAB362; pharmacokinetics; tolerability; safety; ASP8951; immunogenicity
MeSH Terms: conditions — Stomach Neoplasms; Neoplasms | interventions — zolbetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Safety Part Arm A (IMAB362 dose-1/2) (Experimental): Participants will receive a loading dose-1 of IMAB362 on Cycle 1 Day 1 followed by a lower dose-2 in subsequent every 3 weeks.
  Interventions: Drug: Zolbetuximab
- Safety Part Arm B (IMAB362 dose-3) (Experimental): Participants will receive a loading dose-3 of IMAB362 on Day 1 of each cycle (every 3 weeks).
  Interventions: Drug: Zolbetuximab
- Expansion Part (IMAB362 dose-1/2) (Experimental): Participants will receive a loading dose-1 of IMAB362 on Cycle 1 Day 1 followed by a lower dose-2 in subsequent every 3 weeks.
  Interventions: Drug: Zolbetuximab

INTERVENTIONS:
Drug: Zolbetuximab — Zolbetuximab will be administered as a 2-hour intravenous infusion.
  Other Names: IMAB362

SUMMARY:
The purpose of this study is to assess the safety, tolerability and antitumor activity of IMAB362 in Japanese subjects with locally advanced or metastatic Gastric or GEJ adenocarcinoma whose tumors have Claudin (CLDN) 18.2 Expression. This study will also assess pharmacokinetics and immunogenicity of IMAB362.

DETAILED DESCRIPTION:
This study consists of two parts (Part 1: Safety; and Part 2: Expansion). First, the subjects will be enrolled in Safety Part with IMAB362 dose-1/2 (Arm A). Then the safety and tolerability of Arm A will be evaluated at Tolerability Evaluation Meeting (TEM). If there are no safety and tolerability concerns, enrollment for the Safety Part with IMAB362 dose-3 (Arm B) and the Expansion Part with IMAB362 dose-1/2 will be opened. For each part, participants who continue to derive clinical benefit and do not have intolerable toxicity from study treatment will be allowed to remain on treatment until treatment discontinuation criterion is met.

ELIGIBILITY:
Inclusion Criteria:

* Subject has histologically or cytologically confirmed diagnosis of gastric or gastro-esophageal junction adenocarcinoma.
* Subject has gastric or gastroesophageal junction (GEJ) adenocarcinoma based on radiographic imaging or endoscopic examination.
* Subject agrees not to participate in another interventional study while on treatment.
* Subject has Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Subject has predicted life expectancy ≥ 12 weeks.
* Subject must have an available tumor specimen collected at any time prior to the first dose of study treatment.
* Subject must meet all of the pre-specified criteria on the laboratory tests that will be analyzed locally within 7 days prior to the first dose of study drug.
* Locally advanced or Metastatic gastric or GEJ adenocarcinoma with no standard of care treatment option or subject is ineligible to receive available standard of care treatment option.
* Subject's tumor sample has Claudin (CLDN)18.2 membranous staining with any intensity as determined by central Immunohistochemistry (IHC) testing. (Safety part only)
* Subject has CLDN18.2 high expression in ≥75% of tumor cells demonstrating moderate to strong membranous staining as determined by central IHC testing. (Expansion Part Only)
* Subject is an appropriate candidate for a tumor biopsy and is amenable to undergo a tumor biopsy during the Screening period and on-treatment tumor biopsy. (Expansion Part Only)
* Subject has at least 1 measurable lesion according to Response Evaluation Criteria In Solid Tumors (RECIST) 1.1 within 28 days prior to the first dose of study treatment. For subjects with only 1 measurable lesion and prior radiotherapy, the lesion must be outside the field of prior radiotherapy or must have documented progression following radiation therapy. (Expansion Part Only)

Exclusion Criteria:

* Subject has prior severe allergic reaction or intolerance to a monoclonal antibody, including humanized or chimeric antibodies.
* Subject has had radiotherapy within 2 weeks prior to first dose of study drug. Subject who received palliative radiotherapy to peripheral bone metastases within 2 weeks prior to first dose of study drug and has recovered from all acute toxicities is allowed.
* Subject has received other investigational agents or devices concurrently or within 4 weeks prior first dose of study drug.
* Subject has received systemic immunosuppressive therapy, including systemic corticosteroids 2 weeks prior to first dose of study drug. Subjects using a physiologic replacement dose of hydrocortisone or its equivalent are allowed.
* Subject has gastric outlet syndrome or persistent recurrent vomiting.
* Subject has uncontrolled or significant gastrointestinal hemorrhage.
* Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.
* Subject has a known history of a positive test for human immunodeficiency virus (HIV) infection.
* Subject has a positive test for hepatitis B surface antigen (HBsAg) or hepatitis C virus antibody (anti-HCV). Subjects who are negative for HBsAg, but hepatitis B core antibody (HBcAb) positive, hepatitis B virus deoxyribonucleic acid (DNA) test will be performed and if positive will be excluded. Subjects with positive serology but negative HCV ribonucleic acid (RNA) test results are eligible.
* Subject has had within 6 months prior to first dose of study treatment any of the following: unstable angina, myocardial infarction, ventricular arrhythmia requiring intervention or hospitalization for heart failure
* Subject has active infection requiring systemic therapy.
* Subject has clinically significant other disease or co-morbidity, which may adversely affect the safe delivery of treatment within this trial.
* Subject has psychiatric illness or social situations that would preclude study compliance.
* Subject has active autoimmune disease that has required systemic immunosuppressive treatment in the past 2 years.
* Subject has had a major surgical procedure within 28 days prior to the first dose of study drug.
* Subject has Fridericia-corrected QT interval (QTcF) > 450 msec for males and > 470 msec for females on 12-lead electrocardiogram (ECG) at screening based on local testing.
* Subject has any condition which makes the subject unsuitable for study participation.
* Subject has another active malignancy which is likely to require treatment.
* Subjects who find it difficult to adhere to the provisions of treatment and observation specified in the protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2018-06-08 (Actual); Primary Completion 2020-06-09 (Actual); Study Completion 2020-06-09 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicities (DLT) in Safety Part | Up to Day 22
  Any of the IMAB362 related AEs specified as the DLTs will be assessed during the first 3 weeks.
Safety and tolerability assessed by incidence of adverse events (AEs) in Safety Part | Up to 16 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs will be graded using the Common Terminology Criteria for Adverse Events (CTCAE) guidelines (Version 4.03).
Number of participants with laboratory test abnormalities in Safety Part | Up to 14 months
  Number of participants with potentially clinically significant laboratory values will be reported as AEs.
Number of participants with body weight abnormalities in Safety Part | Up to 14 months
  Number of participants with potentially clinically significant body weight change will be reported as AEs.
Number of participants with vital sign abnormalities in Safety Part | Up to 14 months
  Number of participants with potentially clinically significant vital sign values will be reported as AEs.
Number of participants with 12-lead electrocardiogram (ECG) abnormalities in Safety Part | Up to 14 months
  ECGs will be recorded with the participant in the supine position, after the subject has been lying down for approximately 5 minutes. Any clinically significant adverse changes on the ECG will be reported as AEs.
Safety assessed by Eastern Cooperative Oncology Group (ECOG) performance status in Safety Part | Up to 14 months
  Number of participants with potentially clinically significant ECOG performance status values. ECOG grades 0-5, where 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair and 5 = Dead.
Objective Response Rate (ORR) by local review in Expansion Part | Up to 13 months
  ORR is defined as the proportion of participants who have a best overall response of Complete Response (CR) or Partial Response (PR) per Response Evaluation Criteria In Solid Tumors (RECIST) 1.1.

SECONDARY OUTCOMES:
ORR by local review in Safety Part | Up to 13 months
  ORR is defined as the proportion of participants who have a best overall response of CR or PR per RECIST 1.1.
ORR by central review in Expansion Part | Up to 13 months
  ORR is defined as the proportion of participants who have a best overall response of CR or PR per RECIST 1.1.
Disease Control Rate (DCR) in Safety Part and Expansion Part | Up to 13 months
  DCR is defined as the proportion of participants who have a best overall response of CR, PR or stable disease (SD) per RECIST 1.1.
Progression Free Survival (PFS) in Safety Part and Expansion Part | Up to 13 months
  PFS is defined as the time from the date of first dosing until the date of radiological or clinical progressive disease per RECIST 1.1 or death from any cause, whichever is earliest.
Overall Survival (OS) in Safety Part and Expansion Part | Up to 23 months
  OS is defined as the time from the date of randomization until the date of death from any cause.
Duration of Response (DOR) in Safety Part and Expansion Part | Up to 13 months
  DOR is defined as the time from the date of the first response (CR or PR) per RECIST 1.1 to the date of radiological progression or death, whichever occurs earlier.
Pharmacokinetics (PK) of IMAB362 in Safety Part and Expansion Part: Area under the concentration-time curve (AUC) from the time of dosing extrapolated to time infinity (AUCinf) | Up to 3 months
  AUCinf will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Percentage of AUCinf (AUCinf (%extrap)) | Up to 3 months
  AUCinf (%extrap) will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: AUC from the time of dosing to the last measurable concentration (AUClast) | Up to 3 months
  AUClast will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: AUC from the time of dosing to the start of the next dosing interval (AUCtau) | Up to 3 months
  AUCtau will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Maximum concentration (Cmax) | Up to 3 months
  Cmax will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Concentration immediately prior to dosing at multiple dosing (Ctrough) | Up to 16 months
  Ctrough will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Time of the maximum concentration (tmax) | Up to 3 months
  tmax will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Terminal elimination half-life (t1/2) | Up to 3 months
  t1/2 will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Clearance (CL) | Up to 3 months
  CL will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Apparent volume of distribution at steady state (Vss) | Up to 3 months
  Vss will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Apparent volume of distribution during the terminal phase (Vz) | Up to 3 months
  Vz will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Accumulation ratio calculated using AUC (Rac(AUC)) | Up to 3 months
  Rac(AUC) will be derived from the PK serum samples collected.
PK of IMAB362 in Safety Part and Expansion Part: Rac (Cmax) | Up to 3 months
  Rac(Cmax) will be derived from the PK serum samples collected.
Safety assessed by incidence of AEs in Expansion Part | Up to 16 months
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. AEs will be graded using the CTCAE guidelines (Version 4.03).
Number of participants with laboratory test abnormalities in Expansion Part | Up to 14 months
  Number of participants with potentially clinically significant laboratory values will be reported as AEs.
Number of participants with vital sign abnormalities in Expansion Part | Up to 14 months
  Number of participants with potentially clinically significant vital sign values will be reported as AEs.
Number of participants with body weight abnormalities in Expansion Part | Up to 14 months
  Number of participants with potentially clinically significant body weight change will be reported as AEs.
Number of participants with 12-lead ECG abnormalities in Expansion Part | Up to 14 months
  ECGs will be recorded with the participant in the supine position, after the subject has been lying down for approximately 5 minutes. There should be at least 2 minutes between ECG measurements in case a repeat is needed. Any clinically significant adverse changes on the ECG will be reported as AEs.
Safety assessed by ECOG performance status in Expansion Part | Up to 14 months
  Number of participants with potentially clinically significant ECOG performance status values. ECOG grades 0-5, where 0 = Fully active, able to carry on all pre-disease performance without restriction; 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work; 2 = Ambulatory and capable of all self-care but unable to carry out any work activities. Up and about more than 50% of waking hours; 3 = Capable of only limited self-care, confined to bed or chair more than 50% of waking hours; 4 = Completely disabled. Cannot carry on any self-care. Totally confined to bed or chair and 5 = Dead.
Frequency of anti-drug antibody (ADA)-positive participants in Safety Part and Expansion Part | Up to 16 months
  Immunogenicity of IMAB362 will be assessed by the frequency of ADA-positive participants.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (1):
- Site JP00001, Kashiwa, Chiba, Japan

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- [Derived] Shitara K, Xu RH, Ajani JA, Moran D, Guerrero A, Li R, Pavese J, Matsangou M, Bhattacharya P, Ueno Y, Wang X, Shah MA. Global prevalence of claudin 18 isoform 2 in tumors of patients with locally advanced unresectable or metastatic gastric or gastroesophageal junction adenocarcinoma. Gastric Cancer. 2024 Sep;27(5):1058-1068. doi: 10.1007/s10120-024-01518-1. Epub 2024 Jul 2. PMID 38954176
- See also: Link to plain language summary of the study on the Trial Results Summaries website — http://www.trialsummaries.com/Study/StudyDetails?id=25727&tenant=MT_AST_9011